CLINICAL TRIAL: NCT02677883
Title: Manometry- Versus Symptom-Guided Large Volume Thoracentesis: a Randomized Controlled Study
Brief Title: Impact of Pleural Manometry on Chest Discomfort After Therapeutic Thoracentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fabien Maldonado, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VICC THO 1593; NCI-2015-02267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2016-01-18; First posted 2016-02-09 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Manometry-guided thoracentesis (Experimental): Intervention Group - Patients undergo fine needle- aspiration, called therapeutic thoracentesis, to drain fluid accumulated around the lung. Unlike Arm II, the intervention group will have their pleural pressure monitored during the procedure.
  Interventions: Other: Manometry-guided thoracentesis; Other: Symptom-guided thoracentesis
- Arm II: Symptom-guided thoracentesis (Active Comparator): Comparison Group - Patients undergo symptom-guided thoracentesis, the current standard-of-care is to drain fluid until 1) it is all gone or 2) a symptom occurs that indicates the lung may take longer to fully re-expand and drainage should be stopped.
  Interventions: Other: Symptom-guided thoracentesis

INTERVENTIONS:
Other: Manometry-guided thoracentesis — Arm I will undergo a standard of care therapeutic thoracentesis procedure, and in addition include pleural pressure monitoring (via an FDA-approved digital manometer) which is also standard of care but left at the discretion of physicians as per expert recommendations. In this group, the procedure will be stopped when the patient develops symptoms or when all the fluid has been removed, and will also be stopped if the pressure begins to fall quickly in the fluid collection.
  Arms: Arm I: Manometry-guided thoracentesis
Other: Symptom-guided thoracentesis — Arm II will undergo a standard of care therapeutic thoracentesis procedure. In this group, the procedure but will be stopped when the patient develops symptoms or when all the fluid has been removed.

SUMMARY:
This randomized controlled trial attempts to determine whether the measurement of pleural pressures during therapeutic thoracentesis affects the development of chest discomfort after the procedure. During thoracentesis, pleural fluid is drained from the pleural space, resulting in lung expansion. In some cases, the lung is not completely re-expandable, in which case continued drainage results in the development of negative pleural pressures and chest discomfort. Negative pleural pressures may also result in other complications such as re-expansion pulmonary edema and pneumothorax. The identification of negative pleural pressures via manometry during the procedure may lead to a reduction in the complication rate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the impact of pleural manometry on the development of chest discomfort during therapeutic thoracentesis compared to conventional symptom-guided thoracentesis.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo manometry-guided therapeutic thoracentesis.

ARM II: Patients undergo symptom-guided thoracentesis.

ELIGIBILITY:
Inclusion Criteria:

* Referral to pulmonary or interventional radiology services for large-volume thoracentesis
* Presence of a symptomatic moderate or large free-flowing pleural effusion on the basis of:

  * Chest radiograph: effusion filling >= 1/3 the hemithorax, OR
  * Computed tomography (CT)-scan: maximum anteroposterior (AP) depth of the effusion >= 1/3 of the AP dimension on the axial image superior to the hemidiaphragm, including atelectatic lung completely surrounded by effusion, OR
  * Ultrasound: effusion spanning at least three rib spaces with depth of >= 3 cm

Exclusion Criteria:

* Inability to provide informed consent
* Study subject has any disease or condition that interferes with safe completion of the study including:

  * Coagulopathy, with criteria left at the discretion of the operator
  * Hemodynamic instability with systolic blood pressure < 90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the attending physicians
* Pleural effusion is smaller than expected on bedside pre-procedure ultrasound
* Referral is for diagnostic thoracentesis only
* Manometry felt to be clinically indicated
* Inability to assume or maintain a seated position for the procedure
* Presence of multiple loculations on bedside pre-procedure ultrasound

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-26 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Difference in post-procedure chest discomfort scores between control (symptom-guided) and intervention (manometry-guided) groups | one-time assessment, 5 minutes after thoracentesis catheter is removed (on day 1)
  As measured in millimeters along a 10 cm Visual Analog Scale (VAS). The estimated minimal clinically important difference is 15 mm. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention versus (vs) control, will be made using the t-test or Wilcoxon Rank Sum test. Mixed model will be employed to assess the trend of pain score measured across pre-, intra-, and post-procedure.

SECONDARY OUTCOMES:
Change in chest discomfort scores from pre-procedure to post-procedure. | From 1 minute pre-procedure to 5 minutes after thoracentesis catheter is removed (on day 1)
  As measured in millimeters along a 10 cm Visual Analog Scale (VAS). Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention versus (vs) control, will be made using the t-test or Wilcoxon Rank Sum test. Mixed model will be employed to assess the trend of pain score measured across pre-, intra-, and post-procedure.
Incidence of complete lung re-expansion, as assessed by post-procedure chest radiograph | 20 minutes after thoracentesis catheter is removed (on day 1)
  Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Duration of procedure | during the procedure, on day 1, intraoperative
  Measured in seconds, assessed from the time the thoracentesis catheter is introduced to the time the catheter is removed. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the t-test or Wilcoxon Rank Sum test.
Change in subjective report of dyspnea | From 1 minute pre-procedure to 5 minutes after thoracentesis catheter is removed (on day 1)
  Assessed in millimeters along a 10 cm Visual Analog Scale (VAS), from pre-procedure (baseline) to 5 minutes after completion of the procedure. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using either the t-test or Wilcoxon Rank Sum test.
Incidence of clinically-significant re-expansion pulmonary edema | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as present if immediate post-procedure chest radiograph demonstrates new pulmonary edema per radiologist interpretation when compared to pre-procedure radiograph in the hemithorax that underwent thoracentesis, and subject has post-procedure new-onset or worsened hypoxic respiratory failure. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Incidence of pneumothorax | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as either present or absent on the immediate post-procedure chest radiograph per radiologist interpretation. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Incidence of radiographically-apparent re-expansion pulmonary edema | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as present if immediate post-procedure chest radiograph demonstrates new pulmonary edema per radiologist interpretation when compared to pre-procedure radiograph in the hemithorax that underwent thoracentesis. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test
Volume of pleural fluid removed by the thoracentesis procedure | immediately after the thoracentesis catheter is removed, on day 1
  Measured in milliliters. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the t-test or Wilcoxon Rank Sum test.

OTHER OUTCOMES:
Trend in VAS pain scores up to the point at which 1.5L of fluid is removed | at time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Lester M, Maldonado F, Rickman OB, Roller LJ, Avasarala SK, Katsis JM, Lentz RJ. Association between terminal pleural elastance and radiographic lung re-expansion after therapeutic thoracentesis in patients with symptomatic pleural effusion: a post-hoc analysis of a randomised trial. BMJ Open. 2022 Jul 12;12(7):e053606. doi: 10.1136/bmjopen-2021-053606. PMID 35820740
- [Derived] Lentz RJ, Lerner AD, Pannu JK, Merrick CM, Roller L, Walston C, Valenti S, Goddard T, Chen H, Huggins JT, Rickman OB, Yarmus L, Psallidas I, Rahman NM, Light RW, Maldonado F. Routine monitoring with pleural manometry during therapeutic large-volume thoracentesis to prevent pleural-pressure-related complications: a multicentre, single-blind randomised controlled trial. Lancet Respir Med. 2019 May;7(5):447-455. doi: 10.1016/S2213-2600(18)30421-1. Epub 2019 Feb 13. PMID 30772283
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/